CLINICAL TRIAL: NCT03256656
Title: The Effect of Lower Urinary Tract Electrical Stimulation on Renal Urine Production (diuresis) - a Monocentric Basic Study
Brief Title: The Effect of Lower Urinary Tract Electrical Stimulation on Renal Urine Production (diuresis)
Acronym: EFFLUENT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Purpose: Basic Science
Other Study IDs: 2016-01695
Record Dates: First submitted 2017-01-19; First posted 2017-08-22 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Diuresis Under Eletrical Stimulation
MeSH Terms: interventions — Electric Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (2):
- Healthy subjects (Experimental)
  Interventions: Other: electrical stimulation (non painful) of the lower urinary tract to determine the current perception threshold and record sensory evoked potentials
- Patients with SCI (Active Comparator)
  Interventions: Other: electrical stimulation (non painful) of the lower urinary tract to determine the current perception threshold and record sensory evoked potentials

INTERVENTIONS:
Other: electrical stimulation (non painful) of the lower urinary tract to determine the current perception threshold and record sensory evoked potentials

SUMMARY:
In previous studies, in which the perception threshold and / or sensory evoked potentials at different points of the lower urinary tract were examined and measured by means of electrical stimulation, a clear increase in the volume of the bladder and thus the urine excretion under the stimulation could be observed. This observation is now to be investigated more closely in a separate study, in order to strengthen the observation with further measured data and to find possible physiological connections. A detectable influence of electrical stimulation in the lower urinary tract on renal urine production would have a significant relevance both therapeutically and for the neurophysiological understanding of interactions between the lower and upper urinary tracts.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers:

* Written informed consent
* Good mental and physical health
* Age >18 years

Patients with SCI:

* Written informed consent
* Good mental condition
* Age >18 years
* Complete spinal cord injury (AIS A)

Exclusion Criteria:

Healthy volunteers:

* Any neurological or urological pathology
* Pregnancy or breast feeding
* Urinary tract infection (UTI), frequent UTIs
* Hematuria
* Any previous pelvic or spine surgery
* Any craniocerebral surgery
* Any anatomical anomaly of the LUT or genitalia
* Any metabolic disease
* Any renal disease
* Any urinary tract malignancy
* Bladder capacity <150mL or strong desire to void (SDV) already at 60mL

Patients with SCI:

* Any urinary tract malignancy
* Any anatomical anomaly of the LUT or genitalia
* Pregnancy or breast feeding
* Urinary tract infection (UTI), frequent UTIs
* Hematuria
* Any metabolic disease
* Any renal disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2023-10-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in urine output (ml/s) | 10 minutes

SECONDARY OUTCOMES:
Systolic and diastolic blood pressure | Immediately before, during and immediately after the intervention
  Blood pressure is measured using Finometer® device (Finapres Medical Systems, the Netherlands). Unit: mmHg.
Heart rate | Immediately before, during and immediately after the intervention
  Finometer® device (Finapres Medical Systems, the Netherlands). Unit: beats per minute.
Sympathetic skin response | Immediately before, during and immediately after the intervention
  The sympathetic skin response is measured using Finometer® device (Finapres Medical Systems, the Netherlands). Unit: mVs.
Renal restistance index | Immediately before, during and immediately after the intervention
  The resistive index (RI) is measured using Doppler ultrasound
International Consultation on Incontinence Questionnaire-Female Lower Urinary Tract Symptoms (ICIQ-FLUTS) | Once at screening visit
  The ICIQ-FLUTS ("International Consultation on Incontinence Questionnaire Female Lower Urinary Tract Symptoms Module") questionnaire assesses female lower urinary tract symptoms and impact on quality of life. It consists of 12 items covering 3 domains, namely filling symptoms, voiding symptoms and incontinence symptoms. The filling symptoms subscale is the sum of is the sum of item 2 to 5, the voiding symptom subscale is the sum of item 6 to 8 and the incontinence symptoms subscale is the sum of item 9 to 13. The lowest possible score is 0 for all subscales, while the highest possible score is 16 for the filling symptoms subscale, 12 for the voiding symptoms subscale and 20 for the incontinence symptoms subscale. The higher the score, the more symptomatic.
International Consultation on Incontinence Questionnaire-Male Lower Urinary Tract Symptoms (ICIQ-MLUTS) | Once at screening visit
  The ICIQ-MLUTS ("International Consultation on Incontinence Questionnaire Female Lower Urinary Tract Symptoms Module") questionnaire assesses male lower urinary tract symptoms and impact on quality of life. It consists of 13 items covering 2 domains, namely voiding symptoms and incontinence symptoms. The voiding symptoms subscale is the sum of item 2 to 6, while the incontinence symptoms subscale is the sum of item 7-12. The lowest possible score is 0 for both subscales, while the highest possible score is 20 for voiding symptoms subscale and 24 for incontinence symptoms subscale. The higher the score, the more symptomatic
International Prostate Symptom Score (IPSS) | Once at screening visit
  The IPSS ("International Prostate Symptom Questionnaire") score is based on questions concerning urinary symptoms and quality of life (QoL). It consists of 8 items covering 7 urinary symptoms related dimensions (subscales) and 1 additional item assessing quality of life. Each item is rated on a 6-point scale (0=not at all; 5=almost always). The lowest possible score in the total IPSS score is 0 (asymptomatic); the highest possible score is 35 (symptomatic). The QoL index is rated on a 7-point scale, with 0 indicating "delighted" and 6 "terrible."
International Index of Erectile Function (IIEF) questionnaire | Once at screening visit
  The IIEF ("International Index of Erectile Function") is based on questions concerning erectile dysfunction. It consists of 15 items covering 5 domains, namely erectile functioning, orgasmic functioning, sexual desire, and intercourse satisfaction along with a fifth component which encompasses the concept of overall sexual satisfaction. While items 1-10 are rated on a 6-point Likert-type scale from 0 to 5, items 11-15 are rated on a 5-point Likert-type scale from 1 to 5. Higher scores are reflecting less dysfunction. Domain scores are computed by summing the sores for individual items in each domain.
Female Sexual Functioning Index (FSFI) questionnaire | Once at screening visit
  The FSFI ("Female Sexual Function Index") is based on questions concerning female sexual functions. It consists of 19 items covering 6 domains, namely sexual desire, arousal (both subjective and physiologic), lubrication, orgasm, satisfaction, and pain. The lowest possible score in the total FSFI is 2 (asymptomatic); the highest possible score is 36 (symptomatic).
Qualiveen questionnaire | Once at screening visit
  Qualiveen-30 assesses the Specific Impact of Urinary Problems (SIUP) on Quality of Life. It consists of 30 items covering 4 domains, namely inconvenience (9 questions), restrictions (8 questions), fears (8 questions), and impact on daily life (5 questions). Each item is rated on a 5-point ordinal scale (0=asymptomatic; 4=symptomatic). The index of the SIUP on Quality of Life is the mean of the four individual scores. The lowest possible overall score in the Qualiveen-30 is 0 (Urinary problems have no specific impact on QoL); the highest possible score is 30 (Urinary problems have a huge specific impact on QoL).
Lower Urinary Tract Symptoms Quality of Life (LUTS-qol) questionnaire | Once at screening visit
  The LUTS-qol ("International Consultation on Incontinence Questionnaire Lower Urinary Tract Symptoms Quality of Life Module") questionnaire assesses the impact of lower urinary tract symptoms on quality of life. It consists of 20 items. The lowest possible score is 19, while the highest possible score is 76. Greater values are indicating increasing impact on quality of life.
Swiss German Overactive Bladder (OAB) questionnaire | Once at screening visit
  The Swiss German OAB (Swiss German Overactive Bladder) questionnaire assesses to what extent certain bladder symptoms complicated life. It consists of 19 items covering 2 domains, namely symptom bother and health-related quality of life. Each item is rated on an ordinal scale (1-6). The symptom bother score is the sum of item 1 to 6, while the health-related quality of life score is the sum of 13 items. For both domains, the lowest possible score is 0 (no problem), while the highest possible score is 36 for the symptom bother score and 78 for the health-related quality of life score.
Hospital Anxiety and Depression Scale (HADS) questionnaire | Once at screening visit
  The HADS assesses anxiety and depression. It consists of 14 items covering 2 domains, namely anxiety (7 items) and depression (7 items). Each item is rated on an ordinal scale (0-3). An index is separately calculated for the anxiety and depression items. The lowest possible score for anxiety and depression is 0, the highest possible score is 21. A score <8 is considered as normal.
MoCA test | Once at screening visit
  The MoCA ("Montreal Cognitive Assessment") is a screening assessment for detecting cognitive impairment. The lowest possible score is 0, the highest possible score is 31. A score >26 is considered as normal.
Safety outcomes: Incidence of side effects as well as number and intensity/severity (mild/moderate/severe) of adverse events (AE) and serious adverse events (SAE) (Follow-up) | Through study completion until two weeks after last measurement
  Assessed by a 3-day bladder diary
Mean oral fluid intake in mL | Once at screening visit
  Assessed by a 3-day bladder diary
Number of voids per 24 hours | Once at screening visit
  Assessed by a 3-day bladder diary
Number of daytime voids | Once at screening visit
  Assessed by a 3-day bladder diary
Number of nighttime voids | Once at screening visit
  Assessed by a 3-day bladder diary
Number of intermittent catheterizations per 24h | Once at screening visit
  Assessed by a 3-day bladder diary
Number of daytime, intermittent catheterizations per 24h | Once at screening visit
  Assessed by a 3-day bladder diary
Number of nighttime, intermittent catheterizations per 24h | Once at screening visit
  Assessed by a 3-day bladder diary
Mean voided volume in mL | Once at screening visit
  Assessed by a 3-day bladder diary
Mean catheterized post void residual volume in mL | Once at screening visit
  Assessed by a 3-day bladder diary
Pain level score (0 none - 10 worst possible) | Once at screening visit
  Assessed by a 3-day bladder diary
Level of urgency (0 none - 4 severe with incontinence) | Once at screening visit
  Assessed by a 3-day bladder diary
Number of leakages per 24 hours | Once at screening visit
  Assessed by a 3-day bladder diary
Urine leakage (none-heavy) | Once at screening visit
  Assessed by a 3-day bladder diary
Number of used pads per 24 hours | Once at screening visit
  Assessed by a 3-day bladder diary
Wetness of pads (dry-soaked) | Once at screening visit
  Assessed by a 3-day bladder diary

CONTACTS AND LOCATIONS:
Locations (1):
- Balgrist University Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No